CLINICAL TRIAL: NCT01533636
Title: CF And Effects of Drugs Mixed Ex Vivo With Sputum for Mucolytic Treatment to Lung Mucin
Brief Title: CF And Effects of Drugs Mixed Ex Vivo With Sputum for Mucolytic Treatment
Acronym: CADET
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 10-04834
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis, Healthy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of induced and expectorated sputum and blood for DNA and RNA extraction, plasma, and serum will be banked in the UCSF Airway Tissue Bank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: This group will be comprised of healthy individuals without evidence of lung disease.
- Cystic Fibrosis: This group will be comprised of individuals who have been diagnosed with cystic fibrosis.

SUMMARY:
The investigators will collect samples of sputum from healthy volunteers and patients with cystic fibrosis for the purpose of: a) purifying airway mucins for plate-based binding studies and; b) assessment of the effects of carbohydrates on the rheologic properties of the sputum.

This study has two hypotheses:

1. Lectins from Pseudomonas aeruginosa and Aspergillus fumigatus bind to airway mucins in a fucose-dependent manner, and this binding can be inhibited by fucosyl glycomimetic compounds.
2. Fucosyl glycomimetics will compete with Pseudomonas aeruginosa lectin (PA-IIL) and Aspergillus fumigatus lectin (AFL) and disrupt lectin-driven mucin cross-linking in CF sputum.

DETAILED DESCRIPTION:
Pseudomonas lung infection is a major cause of morbidity and mortality occurring in multiple clinical settings. Patients with cystic fibrosis have lung colonization with Pseudomonas from an early age, and overwhelming pseudomonal lung infection is the most common cause of death in these patients. In addition, Pseudomonas pneumonia is common in immunocompromised patients and in patients intubated for management of respiratory failure. Particularly worrisome is the increasing frequency of P. aeruginosa isolates that are resistant to all or most currently available antibiotics. The mechanism of virulence of P. aeruginosa includes soluble lectins that recognize host oligosaccharides on mucins and the cell glycocalyx. P. aeruginosa has two soluble lectins - LecA, also known as PA-IL and LecB, also known as PA-IIL. PA-IL binds galactose and PA-IIL binds fucose. Notably, PA-IIL binds the fucose containing Lewis a oligosaccharide with very high affinity and the role of PA-IIL in biofilm formation is shown by the absence of biofilm formation in Pseudomonas mutants lacking PA-IIL and by the efficacy of multivalent fucosyl-peptide dendrimers in preventing and disrupting Pseudomonas biofilm formation. D-galactose and L-fucose have been successfully used to treat P. aeruginosa infection in a case report, which hints at the potential for glycomimetic therapy in CF. These monosaccharides are weak inhibitors of PA-IIL, however, and multivalent glycomimetics will be needed for more effective inhibition.

Aspergillus fumigatusinfection is responsible for the majority of human and animal aspergillosis disease, even though air sampling studies show that its conidia usually comprise only a small percentage of total airborne fungal challenge. It is both a primary and opportunistic pathogen, and it is particularly troublesome for patients with cystic fibrosis. It causes multiple lung diseases, includingchronic pulmonary aspergillosis, allergic bronchopulmonary aspergillosis, and invasive pulmonary aspergillosis. Aspergillomas also occur in patients with cavitary lung diseases. Together, these diseases cause significant morbidity and mortality, and available treatments are suboptimal. Most patients with chronic pulmonary aspergillosis require antifungal therapy for many months or years, many experience significant drug side effects, and some experience drug resistance. Patients with either allergic bronchopulmonary aspergillosis (ABPA) or severe asthma with fungal sensitization can improve with itraconazole treatment, but relapses are common, and itraconazole affects corticosteroid metabolism and has the potential to worsen steroid side effects. ABPA requires long-term treatment because Aspergillus airway colonization is difficult to eradicate and quickly recurs when treatment is stopped. Immunocompromised patients are especially vulnerable to invasive aspergillosis where the mortality rate is often 50%, even with antifungal treatment. Clearly, therefore, new treatment approaches are needed for lung diseases caused by A. fumigatus, and we are proposing an approach based on prevention of binding to airway mucins. Adherence of A. fumigatus conidia to host tissues has been the subject of extensive research, but little attention has been directed to Aspergillus/mucin interactions, a surprising deficiency given the role mucins play in airway biology.

This study is an ex-vivo study in which we will collect samples of sputum from healthy volunteers and patients with cystic fibrosis for the purpose of: a) purifying airway mucins for plate-based binding studies and; b) ex-vivo assessment of the effects of carbohydrates on the rheologic properties of the sputum.

ELIGIBILITY:
Inclusion Criteria:

* Healthy control subjects:

  * Age 18-65
  * No history of lung disease
* Cystic fibrosis subjects:

  * Age 18-65
  * No history of lung disease other than cystic fibrosis
  * Diagnosis of CF if sweat chloride values > 60 mM on two separate pilocarpine iontophoresis sweat tests and/or two allelic CF-producing mutations in genetic analysis

Exclusion Criteria:

* Use of recreational drugs within 30 days prior to enrollment
* Use of tobacco within 30 days prior to enrollment, or > 10 pack-year tobacco history
* Pregnant or lactating females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cystic Fibrosis and Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2012-07-17 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2026-02-04 (Actual)

PRIMARY OUTCOMES:
Mucus viscosity | Up to one hour

CONTACTS AND LOCATIONS:
Overall Officials: John V Fahy, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- See also: Airway Clinical Research Center website — http://acrc.ucsf.edu